CLINICAL TRIAL: NCT03814122
Title: Examining the Effectiveness of Action-based Cognitive Remediation for First Episode Psychosis
Brief Title: Action-based Cognitive Remediation for First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H2017:214
Record Dates: First submitted 2018-10-12; First posted 2019-01-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cognitive Impairment; Psychosis
MeSH Terms: conditions — Cognitive Dysfunction; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study will be a two-group randomized control cross-over trial. Participants will be randomly assigned to receive ABCR or treatment-as-usual (TAU) for a period of 8 weeks. After this time, the TAU group will receive ABCR. Evaluations of the participant's cognitive functioning, self-esteem, psychotic symptoms, and functional skills will be completed at baseline, post-treatment (approximately 8 weeks), and 16 weeks later.
Who Masked: Outcomes Assessor
Masking Description: Pre- and post- assessments will be administered by someone blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABCR Treatment Group (Experimental): Group that is immediately administered action-based cognitive remediation intervention.
  Interventions: Behavioral: Action-based cognitive remediation
- Waitlist Control Group (Active Comparator): Group that is waitlisted (i.e., receives treatment-as-usual) and after approximately 8 weeks received action-based cognitive remediation intervention
  Interventions: Behavioral: Action-based cognitive remediation; Other: Waitlist Control Group

INTERVENTIONS:
Behavioral: Action-based cognitive remediation — Action-Based Cognitive Remediation (ABCR) is a new program that was developed to address the challenges of transferring cognitive gains to improved quality of life and reduced disability. ABCR combines traditional cognitive training with an added behavioural component (e.g., role-plays, simulations of real world tasks) to foster learning through rehearsal and procedural memory which increases the likelihood of participants bridging cognitive strategies into real-world activities. ABCR also includes goal setting and behavioural activation procedures to stimulate transfer of in-session gains to everyday life changes.
Other: Waitlist Control Group — Receive treatment-as-usual through regular early psychosis programming.
  Arms: Waitlist Control Group

SUMMARY:
Cognitive impairments are a core and enduring feature of first-episode psychosis and schizophrenia, and are associated with significant functional impairment. Cognitive remediation (CR) is a behavioural intervention that has been found to have a small to moderate effect on cognition in individuals with schizophrenia, and recent studies suggests that it leads to improved cognition in persons with first-episode psychosis. Results from a CR feasibility project that was conducted through the Winnipeg Regional Health Authority's Early Psychosis Prevention and Intervention Service (EPPIS) showed promising findings. Specifically, large effect sizes were found in the areas of verbal learning and self-esteem. Moreover, the intervention was found to be acceptable to the participants. However, the findings are limited by the sample size and lack of control group.

In this proposed study, the investigators seek to expand the scientific support for treating neurocognitive impairments in order to increase functional productivity associated with first-episode psychosis. A novel group CR program, action-based cognitive remediation (ABCR), has been developed by Dr. C. Bowie (co-investigator) to promote the generalization of cognitive skills to real-world activities. ABCR has been found to improve both cognition and functional competence in persons with schizophrenia. The primary outcome measure will examine whether ABCR results in improved executive functioning in persons with first-episode psychosis compared to psychiatric rehabilitation alone. Secondary outcome measures (e.g., memory, processing speed, self-esteem, emotional functioning, adaptive functioning) will also be analyzed.

DETAILED DESCRIPTION:
The proposed study will be a two-group randomized control cross-over trial. Participants will be recruited from EPPIS and will be randomly assigned to receive ABCR or treatment-as-usual (TAU) for a period of 8 weeks. After this time, the TAU group will receive ABCR. TAU will be the psychiatric rehabilitation programming offered to all patients enrolled with EPPIS. ABCR will consist of two, 2-hour groups/week, for a period of 8 weeks. Each group session will consist of: (1) computerized cognitive training using Scientific Brain Training Pro (an online program used in previous CR and ABCR research), (2) strategic monitoring (i.e., increasing awareness of cognitive strategies used and learning to switch strategies as needed), (3) role-plays and simulations of real world tasks to facilitate the transfer of skills to functioning, and (4) goal setting and cognitive approach planning. ABCR builds on procedural learning skills with explicit work-related role-plays to facilitate the immediate and salient abstraction of drill and practice remediation techniques. The activities are work skills that were developed by Dr. Bowie (co-investigator) in collaboration with community vocational rehabilitation partners. The props match those used in work settings and were designed on a miniature scale and include a cash register, filing system, conveyer belt, cleaning closet, garden nursery, and secretarial station. The activities in ABCR capitalize on procedural learning skills through role-plays and props that simulate a work environment. In ABCR, the important aspects of drill and practice, strategic monitoring to enhance flexible problem solving approaches, and bridging are maintained. The role-plays immediately follow the computerized drill and practice exercise and therapists facilitate group discussions of how the cognitive skills and flexibility in thinking from drill and practice can be effective while directly engaged in an everyday work environment. Thus, the bridging used in ABCR is a tangible, procedural, and realistic. This approach to bridging differentiates the treatment from standard CR, where the discussion-based approach is limited by the auditory learning, memory, and abstraction deficits typically observed in psychosis. ABCR group sessions will be facilitated by the Primary Investigator and trained bachelor's or master's level research assistants/psychology residents who will be trained and supervised by the Primary Investigator. Participants will also be encouraged to complete computerized cognitive training using the online program, Scientific Brain Training Pro as supplemental homework exercises outside of the scheduled treatment group (20 minutes/day). Due to the online nature of this program, participants can access this program either at their personal homes or at EPPIS.

Evaluations of each participant's cognitive functioning, self-esteem, psychotic symptoms, and functional skills will be completed at baseline and post-treatment (approximately 8 weeks later). The TAU group will then participate in ABCR and all participants will be re-evaluated following completion of the second intervention (at approximately 16 weeks post-baseline). Testing will be administered by trained bachelor's or master's level research assistants who are blind to study hypothesis or group assignment. These assistants will be trained and supervised by the Primary Investigator. Test batteries will be presented in counterbalanced order and, when possible, alternate forms will be used to reduce the likelihood of practice effects.Using a repeated measures analysis of covariance (ANCOVA), the treatment and control group's post-intervention data will be compared while controlling for pre-treatment scores. For all analyses, p < .05 will be used as the statistical threshold for significance.

ELIGIBILITY:
Inclusion Criteria:

* Involved in the Winnipeg Regional Health Authority's Early Psychosis Prevention and Intervention Service
* Must be at least 18 years old
* Be proficient in English
* Have stable medication orders for 3 months
* Have capacity to voluntarily consent to participate in the treatment study

Exclusion Criteria:

* Organic brain damage
* Intellectual disability

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Executive Functioning; Wisconsin Card Sorting Test (Heaton and PAR Staff, 2005). | Baseline, after approximately 8 weeks and 16 weeks
  Commonly used neuropsychological computerized test to assess the ability to form abstract concepts, to shift and maintain set, and to utilize feedback. Total number of categories completed and perseverative errors (reported as t-score with range <20 to >80) will be reported. Higher values indicate better outcome. More information can be found at: http://www4.parinc.com/Products/Product.aspx?ProductID=WCST

SECONDARY OUTCOMES:
Change in Cognitive Functioning; Screen for Cognitive Impairment in Psychiatry (Purdon, 2005). | Baseline, after approximately 8 weeks and 16 weeks
  Scale for screening cognitive deficits in persons with schizophrenia and psychiatry, including verbal learning and memory, auditory working memory, verbal fluency and visuomotor tracking. Total score reported as a z-score (range of -3 to +3). Higher values indicate better performance.
Change in Psychotic Symptoms; Brief Psychotic Rating Scale (Overall & Gorham, 1962). | Baseline, after approximately 8 weeks and 16 weeks
  A 24-item measure commonly used in research and clinical settings that is designed to quantify the severity of positive and negative symptoms of psychosis. Scale ranges from 24-168. Higher values indicate greater number and severity of symptoms.
Change in Functional Skills; Canadian Objective Life Skills (COALS) (McDermid Vaz & Heinrichs) | Baseline, after approximately 8 weeks and 16 weeks
  Participants are examined with a series of role-playing tasks for their comprehension and planning of recreational activities, financial skills in handling money and writing checks, use of a telephone for instrumental communication, and ability to use information from bus schedules and maps to use public transportation effectively. Total score ranges from 0-60. Higher value indicates better performance.
Change in Visual Memory; Brief visuospatial memory test-revised (Benedict, 1997). | Baseline, after approximately 8 weeks and 16 weeks
  Commonly-used neuropsychological measure of visual learning and memory that uses a multiple-figural test to assess immediate memory, delayed memory and recognition abilities. Recall scores are reported as t-scores (range: <20-80) and higher values indicate better performance. Please note that a copy of the test protocol cannot be provided due to copyright protection, but more information can be found at: http://www4.parinc.com/Products/Product.aspx?ProductID=BVMT.
Change in Self-Esteem; Rosenberg Self-Esteem Scale (Rosenberg, 1965). | Baseline, after approximately 8 weeks and 16 weeks
  A 10-item measure that is commonly used to measure self-esteem. Respondents are asked to read a list of statements dealing with general feelings about themselves and rate each one on a four-point scale from SD =Strongly Disagree (score of 0) to SA =Strongly Agree (score of 3). Scores are summed to provide a total score for the measure. Total score ranges from 0-30, with higher values indicating higher self-esteem.
Change in Disability Beliefs; World Health Organization Disability Assessment Schedule II (World Health Organization) | Baseline, after approximately 8 weeks and 16 weeks
  36-item self-administered measure that assesses disability in adults over 18 years. Total score ranges from 0-144 with higher scores indicating greater perceived disability.
Change in Illness Beliefs; Personal Beliefs About Illness Questionnaire-Revised (Birchwood, Jackson, Brunet, Holden & Barton, 2012). | Baseline, after approximately 8 weeks and 16 weeks
  20-item, self-report measure that assesses common psychological reactions related to loss, social marginalization, shame, entrapment, and control in persons with a first-episode psychosis. Total score ranges from 0-60. Higher scores indicate negative reactions to the diagnosis.
Change in Perceived Competence; Perceived Competence for Learning Scale | Baseline, after approximately 8 weeks and 16 weeks
  4-item self-report measure assessing person's feeling of competence to master learning material. Total score ranges from 4-28. Higher scores indicate greater perceived competence.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Murphy, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Crisis Response Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No